CLINICAL TRIAL: NCT01669603
Title: Effect of Probiotic on the Innate and Adaptive Host Response to Rhinovirus (EPIARR)
Acronym: EPIARR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Principal Investigator, Ronald Turner, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16241
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Common Cold
Keywords: Common cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacterium animalis lactis Bl-04 (Experimental): Bifidobacterium animalis subspecies lactis Bl-04 as powder mixed into drink.
  Interventions: Dietary Supplement: Bifidobacterium lactis Bl-04; Biological: Rhinovirus
- Placebo (Placebo Comparator): Placebo will be 1g of sucrose that has identical appearance, smell, and taste with the study product.
  Interventions: Dietary Supplement: Placebo; Biological: Rhinovirus

INTERVENTIONS:
Dietary Supplement: Bifidobacterium lactis Bl-04 — The study product will be a 2*109 cfus of probiotic Bifidobacterium lactis Bl-04 mixed with 1g of sucrose as a carrier.
  Arms: Bifidobacterium animalis lactis Bl-04
Dietary Supplement: Placebo — Placebo will be 1g of sucrose that has identical appearance, smell, and taste with the study product.
  Arms: Placebo
Biological: Rhinovirus — rhinovirus for experimental challenge

SUMMARY:
The study is designed to assess the effect of ingestion of a probiotic on innate and adaptive host responses to rhinovirus infection.

DETAILED DESCRIPTION:
The common cold is a ubiquitous illness of man that is associated with significant medical and socioeconomic consequences. Current treatments for the common cold that have proven efficacy are limited to pharmacologic agents that are directed at specific symptoms. These treatments- antihistamines, nasal decongestants and analgesics- have limited effectiveness, generally relieving the target symptom by 15-25% at the peak of activity, and are associated with bothersome side effects. There are no currently effective treatments for prevention of rhinovirus infections.

Probiotics have been defined by FAO/WHO as "Live microorganisms which when administered in adequate amount confer a health benefit on a host." The most common probiotics belong to Lactobacillus or Bifidobacterium genera. Bifidobacteria are natural human gut inhabitants that were discovered over a hundred years ago from the feces of breast-fed infants. The study product Bifidobacterium animalis subspecies (subsp.) lactis Bl-04 (Bl-04) has been genetically characterized as B. animalis subsp. lactis by 16S rRNA gene sequencing and full genome sequence comparison. Bl-04 has been deposited in the American Type Culture Collections safe deposit as SD5219.

This study will test the hypothesis that ingestion of a probiotic Bifidobacterium animalis subsp. lactis Bl-04 will alter the innate and adaptive host response to rhinovirus infection.

ELIGIBILITY:
Inclusion Criteria:

AT ENROLLMENT:

* Subject must be 18-60 years of age.
* Subject must read and sign a copy of the approved Consent Form
* Female subjects must be using an effective birth control method.

INCLUSION CRITERIA AT DAY -28

* Subject must read and sign a copy of the approved Consent Form

AT CHALLENGE:

* Female subjects must be using an effective birth control method.
* Subject must have a serum neutralizing antibody titer of less than or equal to 1:4 to rhinovirus type 39

Exclusion Criteria:

AT ENROLLMENT:

* Current cancer diagnosis or immunosuppressive therapy in the last 6 months
* Any clinically significant abnormalities of the upper respiratory tract
* Any clinically significant acute or chronic respiratory illness
* Any clinically significant bleeding tendency by history
* Hypertension that requires treatment with antihypertensive medications
* History of angina or other clinically significant cardiac disease
* Any medical condition that in the opinion of the Principal Investigator is cause for exclusion from the study
* History of regular use (more than 3 days in 7) of tobacco products within the preceding two weeks
* History of drug or alcohol abuse in the 6 months preceding the study

EXCLUSION CRITERIA AT DAY -28

* Antibiotic use within 3 months prior to study start
* Female subjects with a positive urine pregnancy screen.
* History of use of probiotics in the preceding 2 weeks.

EXCLUSION CRITERIA AT CHALLENGE:

* Any upper respiratory infection or allergic rhinitis in the two weeks prior to the start of the study
* Any medical condition that in the opinion of the Principal Investigator is cause for exclusion from the study
* Use of any anti-inflammatory (steroids or NSAIDs) or cough/cold preparation in the two weeks prior to the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 789 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Turner, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Turner RB, Woodfolk JA, Borish L, Steinke JW, Patrie JT, Muehling LM, Lahtinen S, Lehtinen MJ. Effect of probiotic on innate inflammatory response and viral shedding in experimental rhinovirus infection - a randomised controlled trial. Benef Microbes. 2017 Apr 26;8(2):207-215. doi: 10.3920/BM2016.0160. Epub 2017 Mar 27. PMID 28343401

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 789 subjects were screened for participation. 190 subjects met all study criteria for randomization to study intervention.
Period: Overall Study
Arm/Group | Bifidobacterium Animalis Lactis Bl-04 | Placebo
Started | 95 | 95
Completed | 58 | 57
Not Completed | 37 | 38

BASELINE CHARACTERISTICS:
Population: Volunteers challenged with rhinovirus who met protocol definitions for analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bifidobacterium Animalis Lactis Bl-04 | Placebo | Total
Number analyzed (Participants) | 95 | 95 | 190
Age, Categorical [Count of Participants; unit: Participants] — Population: Analysis limited to participants who were susceptible to RV39, had no virus detected in nasal lavage on Day 0, were infected and completed the study.
  Participants
    number analyzed (Participants) | 58 | 57 | 115
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 58 | 57 | 115
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: analysis cohort was those volunteers who were susceptible to RV-A39 by neutralizing antibody titer, had no virus detected in the nasal lavage on day 0, and who were infected and completed the study
  years
    number analyzed (Participants) | 58 | 57 | 115
    (all) | 22 (6) | 23 (7) | 23 (7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: analysis cohort was those volunteers who were susceptible to RV-A39 by neutralizing antibody titer, had no virus detected in the nasal lavage on day 0, and who were infected and completed the study
  Participants
    number analyzed (Participants) | 58 | 57 | 115
    Female | 39 | 33 | 72
    Male | 19 | 24 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: analysis cohort was those volunteers who were susceptible to RV-A39 by neutralizing antibody titer, had no virus detected in the nasal lavage on day 0, and who were infected and completed the study
  Participants
    number analyzed (Participants) | 58 | 57 | 115
    Hispanic or Latino | 3 | 4 | 7
    Not Hispanic or Latino | 54 | 52 | 106
    Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: analysis cohort was those volunteers who were susceptible to RV-A39 by neutralizing antibody titer, had no virus detected in the nasal lavage on day 0, and who were infected and completed the study
  Participants
    number analyzed (Participants) | 58 | 57 | 115
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 8 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 2 | 5
    White | 52 | 46 | 98
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 95 | 95 | 190

OUTCOME MEASURES:

1. Primary Outcome: Interleukin-8 (IL-8)
Description: Nasal lavage will be performed to collect and measure IL-8.
Time Frame: 72 hours
Population: analysis cohort was those volunteers who were susceptible to RV-A39 by neutralizing antibody titer, had no virus detected in the nasal lavage on day 0, and who were infected and completed the study
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Arm/Group | Bifidobacterium Animalis Lactis Bl-04 | Placebo
Number analyzed (Participants) | 58 | 57
pg/ml | 133 (2.5) | 122 (2.9)

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Bifidobacterium Animalis Lactis Bl-04 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/95
Other Adverse Events (participants affected / at risk) | 4/95 | 1/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bifidobacterium Animalis Lactis Bl-04 (N=95) | Placebo (N=95)
gastrointestinal (Gastrointestinal disorders) | 4 (4) | 0 (0)
respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No